CLINICAL TRIAL: NCT06069739
Title: Development and Evaluation of a Health Education Programme Through Physical Exercise for the Development of Autonomous Physical Activity Habits in People With Severe Mental Disorders
Brief Title: Health Education Programme Through Physical Exercise for People With Severe Mental Disorders
Acronym: HEPPE-PSMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physical exercise programme
Record Dates: First submitted 2023-09-05; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Severe Mental Disorder; Obesity
Keywords: Exercise; Neurocognition; Inflammation; Oxidative stress; Vascular damage; Metabolic activity; Mental illnesses; Obesity
MeSH Terms: conditions — Mental Disorders; Obesity; Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: Eligible participants were randomly assigned in a 1:1 ratio to a 12-week program of either; (a) guided-exercise of moderate intensity and frecuency, and incentive of autonomous physical activity proposals by the specialist; guided physical activity group (GPAG), or (b) 12 weeks of an exercise program standard physical activity without guided and incentives; standard physical activity group (SPAG). Both groups followed the same randomized recruitment procedure, data collection and follow-up. All treatment sessions were conducted from March to June 2016. To maintain the rigor of the research, possible risks that could question the internal and external validity of the study results were identified and strategies were proposed to eliminate them.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided physical activity group (Experimental): Guided-exercise of moderate intensity and frecuency, and incentive of autonomous physical activity proposals by the specialist.
  Interventions: Behavioral: Guided physical activity
- Standard physical activity group (Active Comparator): Standard physical activity without guided and incentives.
  Interventions: Behavioral: Standard physical activity

INTERVENTIONS:
Behavioral: Guided physical activity — To achieve the European guidelines of 150 minutes by week of moderate intensity physical activity, participants randomized to the GPAG condition were prescribed three 60 minutes exercise sessions (five minutes of warm-up and five minutes of cool-down for a total of sixty minutes per session) per week for 12 weeks. Exercise consisted of brisk walking in urban and rural open spaces during which heart rate monitors were worn and participants were instructed to stay within their moderate intensity range. The incentives were different proposals for specific exercises to train the different musculoskeletal areas more comprehensively. Autonomous exercise was monitored offside the sessions through a series of weekly checkpoints.
  Arms: Guided physical activity group
Behavioral: Standard physical activity — Participants randomised to the SPAG performed their usual daily activities and continued with their daily routine.
  Both conditions were matched for duration of physical activity. Participants in both conditions were required to attend three on-site sessions by week over 12 weeks that served as checkpoints. Moreover, both conditions were provided with brief healthy lifestyle counseling at baseline.
  Arms: Standard physical activity group

SUMMARY:
The goal of this clinical trial is to [learn about, test, compare etc.] in individuals with severe mental disorders and obesity comorbid.

The main question[s] it aims to answer are:

* Are inflammatory activity, oxidative and vascular damage and metabolic mechanisms, as well as neurocognitive and functional performance, related to different physical exercise interventions?
* Do inflammatory, oxidative stress and cardiometabolic biomarkers predict neurocognitive improvement after physical activity training?

Participants will guided-exercise of moderate intensity and frecuency, and incentive of autonomous physical activity proposals by the specialist; guided physical activity group (GPAG), or (b) 12 weeks of an exercise program standard physical activity without guided and incentives; standard physical activity group (SPAG).

If there is a comparison group: Researchers will compare GPAG and SPAG to see if inflammatory, oxidative stress, and cardio-metabolic biomarkers improve neurocognitive performance after physical activity training

DETAILED DESCRIPTION:
The psychiatric disorders and obesity comorbidity is related to neurocognitive impairment and inflammation. Exercise is crucial to improve and maintain healthy lifestyles. This randomized controlled trial tested the efficacy of aerobic exercise as promoter of neurocognitive improvement across psychiatric disorders and OB comorbid. Participants (n=29) received brief healthy lifestyle counseling and were randomized to 12 weeks of guided-exercise of moderate intensity and frequency, and incentive of autonomous physical activity proposals by the specialist; guided physical activity group (GPAG) (n=10) or 12 weeks of exercise standard physical activity without guided and incentives; standard physical activity group (SPAG) (n=19). Peripheral blood biomarkers of inflammation, oxidative stress, vascular mechanisms and metabolic activity, as well as neurocognitive and functional performance were assessed twice over after and before treatment. Mixed one-way analysis of variance and linear regression analyses were performed.

ELIGIBILITY:
Inclusion Criteria:

* MDD, BD and SZ were diagnosed according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders - DSM-5 (APA, 2014).
* Participants with MDD and BD should meet the remission criteria (Tohen et al., 2009) of an acute affective episode, defined as Young Mania Rating Scale (YMRS) score ≤ 6 and Hamilton Rating Scale for Depression (HRSD) score ≤ 8, and individuals with SZ had to be clinically stable, defined as Positive and Negative Syndrome Scale (PANSS) score ≤ 36.
* The comorbid OB diagnosis was based on World Health Organization (WHO) criteria.
* Ability to understand study procedures and willingness to give written consent was required for participation.

For recruitment as HC

* Absence of physical illness
* Absence of pharmacological treatments
* Absence of family history of psychiatric disorders in first-degree relatives were required.
* Ability to understand study procedures and willingness to give written consent was required for participation.

Exclusion Criteria:

* current hospitalization
* documented cognitive impairment not secondary to psychiatric disorder (intellectual disability or major neurocognitive disorder, i.e. dementia)
* disability or inability that prevented understanding of the protocol
* current substance use disorders (except for nicotine)
* pregnancy
* intake of steroids
* corticosteroids, antioxidants, antibiotics, and immunologic therapies
* fever over 38°C
* history of vaccination within 4 weeks of the evaluation
* medical contraindications for exercise
* body mass index ≥ 40
* diastolic/systolic blood pressure ≥ 140/90
* resting heart rate ≥ 100.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Verbal learning and memory | 4 months
  Complutense Verbal Learning Test total immediate recall, short-term free recall and long-term free recall The higher scores mean a better outcome.
Cognitive flexibility | 4 months
  Wisconsin Card Sorting Test The higher scores mean a better outcome.
Verbal fluency | 4 months
  Animal naming test for phonemic and semantic fluency. The higher scores mean a better outcome.
Working memory | 4 months
  Trail Making Test The higher scores mean a better outcome.
Short-term memory | 4 months
  Complutense Verbal Learning Test total immediate recall, short-term free recall and long-term free recall The higher scores mean a better outcome.
Visual memory | 4 months
  Rey-Osterrieth Complex Figure Test figure two minutes after the copy and 20 minutes after the copy.
  The higher scores mean a better outcome.
Processing speed | 4 months
  Stroop Color and Word test color/word subtest The higher scores mean a better outcome.
Functional Assessment Short Test | 4 months
  Functional performance. The higher scores mean a better outcome.
Short Form-36 Health Survey questionnaire | 4 months
  Quality of life. The higher scores mean a better outcome.
World Health Organization Quality of Life brief scale | 4 months
  Quality of life. The higher scores mean a better outcome.
Inflammatory markers | 4 months
  Serum cytokine concentrations were determined using Luminex® X-MAP technology (Luminex Corp., Austin, TX, USA) based on flow cytometry. Sample processing and data analysis were performed according to the manufacturer's instructions. (Behring Nephelometer II, Dade Behring, Inc., Newark, DE, USA)..
Oxidative stress markers | 4 months
  Oxidative stress in leukocytes was evaluated using fluorimetry techniques with a fluoroscan (Synergy MX). In total, 100 000 cells were plated in each well of 96-well plates and incubated for 30 min at 37 °C with the corresponding fluorochromes, as follows: dichlorofluorescein diacetate to measure reactive oxygen species (ROS) production (485 nm excitation, 535 nm emission), MitoSOX to measure mitochondrial ROS (mROS) (510 nm excitation, 580 nm emission), tetramethylrodamin methyl ester to assess mitochondrial membrane potential (552 nm excitation, 574 nm emission), nonylacridin orange mitochondrial mass (495 nm excitation, 519 nm emission), and 5-chloromethylfluorescein diacetate to measure intracellular glutathione (492 nm excitation, 517 nm emission). The monocyte cell line U-937 was used as an internal control to avoid potential fluctuations in fluorescence over time.
Adhesion molecules markers | 4 months
  Serum lipid peroxidation levels were measured using a commercial thiobarbituric acid reactive substances (TBARS) kit according to the manufacturer's instructions (Olympus, Hamburg, Germany). A Luminex 200 flow analyzer system (Austin, TX, USA) was employed to analyze adhesion molecules in serum. To measure immunological markers, citrated blood samples were incubated with dextran (3%) for 45 min to isolate human polymorphonuclear leukocytes (PMNs). The supernatant was layered over Ficoll-Hypaque (GE Healthcare, Barcelona, Spain) and centrifuged for 25 min at room temperature at 650g. Lysis buffer was added to the remaining erythrocytes in the pellet, which were incubated at room temperature for 5 min and then spun at 240g for 5 min. PMNs were rinsed twice and resuspended at 37 ℃ in Hanks' balanced salt solution (Sigma Aldrich, MO). Scepter 2.0 cell counters (Millipore, MA, USA) was employed to count cells
Metabolic markers | 4 months
  Under aseptic conditions, fasting venous blood samples were collected between 8 and 9 am to measure.
Maximum heart rate | 4 months
  Measured with a watch-shaped device that was worn on the wrist and captured the beats per minute.
Systolic pressure/diastolic pressure | 4 months
  Measured on the right arm using an automatic sphygmomanometer with participants in the sitting position after resting for 5 minutes.
Waist circumference | 4 months
  Measured in the standing position at the end of normal expiration and at the midway between the inferior costal margin and the superior border of the iliac crest.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Tabarés-Seisdedos, Principal Investigator — Consorcio Centro de Investigación Biomédica en Red (CIBER)

IPD SHARING:
Plan to Share IPD: No